CLINICAL TRIAL: NCT05788796
Title: The Effect of Band-Aid Applied to the Umbilical Area on Nausea and Vomiting During Pregnancy
Brief Title: The Effect of Plaster on Nausea-Vomiting During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, : Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13.03.2023
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Nausea Gravidarum; Vomiting of Pregnancy; Pregnancy Related; Acupressure
Keywords: Pregnancy; Nausea; Vomiting; Acupressure
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Pregnant women in the application group will be asked to take a hazelnut-sized cotton ball before going to bed, put it in the middle of the navel and close it diagonally with a band-aid.
  Pregnant women in the control group will be asked not to make any lifestyle changes and to continue their routine daily lives.
Masking Description: Since there is no placebo group, masking will not be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Experimental group (Experimental): Experimental:Pregnant women in the application group will be asked to take a hazelnut-sized cotton ball before going to bed, put it in the middle of the navel and close it diagonally with a band-aid.
  Interventions: Behavioral: Band-aid application
- Assigned Interventions (No Intervention): No Intervention: Control group Pregnant women in the control group will be asked not to make any lifestyle changes and to continue their routine daily lives.

INTERVENTIONS:
Behavioral: Band-aid application — Before starting the study, cotton and band-aids will be provided to the women in the application group by the researchers.
  • Pregnant women in the application group will be asked to take a hazelnut-sized cotton ball before going to bed, put it in the middle of the navel and close it diagonally with a band-aid.
  Arms: Experimental: Experimental group

SUMMARY:
Hormonal and physical changes during pregnancy can cause nausea and vomiting. Nausea and vomiting are common, especially in the first trimester. The incidence of nausea and vomiting during pregnancy varies between 50% and 80%. Symptoms range from mild nausea to excessive vomiting, dehydration, electrolyte imbalances, and weight loss to a severe form of nausea-vomiting called hyperemesis gravidarum (HG). Nausea-vomiting can cause discomfort in the pregnant woman in its mildest form, and a serious threat to the life of the mother and fetus in the most severe form. Nausea and vomiting during pregnancy is an important symptom that reduces the quality of life of the pregnant woman.In order to reduce the complaints of nausea and vomiting during pregnancy, women are offered suggestions such as changing their eating habits and staying away from stress. Complementary and alternative methods can also be used to reduce nausea and vomiting. Acupressure, which is one of these methods, is accepted as an important, effective, supportive and economical complementary method as a non-invasive technique that midwives can directly include in the control of nausea and vomiting during pregnancy, reducing the severity of labor pain, accelerating the birth process, gynecological problems and assisting breastfeeding. The efficacy of acupressure applied to P6, ST36 and CV8 points in cases of nausea and vomiting experienced after motion sickness, chemotherapy or surgery has been investigated in many studies. The CV8 point has not been studied sufficiently in reducing nausea and vomiting in pregnancy. Therefore, the aim of this study is to investigate the effect of a band-aid applied to the umbilical area (Shenque-CV8 point), which is a method that pregnant women can apply on their own, on nausea-vomiting during pregnancy.The sample of the study will consist of 60 pregnant women, 30 in the application group and 30 in the control group. Which of the application/control groups of the pregnant women constituting the sample group will be included will be determined by simple randomization. Pregnant women in the treatment group will be asked to fix a hazelnut-sized cotton ball to their navel with a Band-Aid regularly for five days before going to bed at night. Pregnant women in the control group will not be asked to make any life changes. Five days later, the nausea-vomiting levels of the pregnant women who applied and the pregnant women in the control group will be compared.

DETAILED DESCRIPTION:
Pregnancy is a process that affects life more or less as a result of hormonal, physical and psychological changes in the woman's body (Bustos et al. 2017; Karataş and Mete 2012). For this reason, the changes that occur during pregnancy can sometimes lead to deterioration of the general health status and unexpected problems. In order for the pregnancy to continue and result in a healthy way, the physical and mental safety of the pregnant must be ensured (Bustos et al. 2017). One of the most common problems experienced by women during pregnancy is early pregnancy nausea and vomiting, the cause of which is not yet known and affects 50-80% of pregnant women (Laitinen 2020, Şimşek 2021). Nausea and vomiting in pregnancy usually begin in the early weeks of pregnancy and disappear spontaneously at the beginning of the second trimester. However, in some cases, a more severe picture called hyperemesis gravidarum may be seen, which may require hospitalization and accompanied by conditions such as weight loss and fluid-electrolyte imbalance (Özdemir et al, 2010; Lee and Saha, 2011). Pregnancy hormones (hCG, estradiol, progesterone), upper gastrointestinal system (GIS) disorders, Helicobacter pylori, hyperthyroidism, immune system and nutritional disorders and psychological factors are among the factors thought to cause nausea and vomiting during pregnancy (Bustos et al. 2017; Timur and Kızılırmak 2011; Aşcı and Özer 2011).The prevalence of nausea in pregnancy is 50-80% (Einarson et al. 2013; Pepe and Ege 2019; Mutlugüneş and Mete 2019), while the prevalence of vomiting and retching is 50% (Matthews et al. 2015). Nausea-vomiting is usually time-limited and starts at the 5th week of pregnancy (Gürbüz and Güngör 2018), 8-12. It peaks in the 14th week and decreases after the 14th week, in some cases 16-18. It can last up to weeks (Bustos et al. 2017; Timur and Kızılırmak 2011; Matthews et al. 2015; Özdemir et al. 2010). The probability of recurrence in the next pregnancies of women is 15-81% (Musfirowati et al. 2018; ACOG 2018).Not knowing when nausea and vomiting will end and how to manage it causes emotional disappointment, hopelessness, weakness and anxiety in pregnant women. This prevents the pregnant woman from coping with nausea and vomiting, and makes it difficult to adapt to pregnancy and motherhood afterwards (Mete et al. 2009). Since its etiology is multifactorial, symptomatic treatment is applied to cope with nausea and vomiting. Pregnant women mostly do not prefer drug treatment because of the possibility of adversely affecting the fetus and give more priority to non-drug methods (Timur and Kızılırmak 2011). In the literature, it is stated that people tend to use non-drug methods such as hypnotherapy, behavioral therapy, regulation of nutrition and life routines, massage, acupuncture and herbal treatments to control nausea and vomiting (Aşcı and Özer 2011; Heuvel et al. 2016; Mohammadbeıgı et al. 2011). ; Viljoen et al. 2014; Kia et al. 2014). Acupressure is also one of the non-drug methods. In terms of ease of application and effectiveness, acupressure emerges as a method used in the control of symptoms in different diseases (Çalık and Kömürcü 2014). acupressure; It is a treatment method applied to points in certain parts of the body with finger pressure or a band that can make this pressure.The difference of the acupressure method from acupuncture is that by applying pressure to certain points with the fingers and the palm of the hand instead of the needle, the energy density collected in the region is distributed and the organs associated with the relevant points are relieved in this way (Çalık and Kömürcü 2014; Arslan and Özdemir 2015). Acupressure method; it is an easy-to-apply, economical, and side-effect-free method (Lee et al. 2008). Acupressure points used in cases such as nausea-vomiting; P6 (Pericardium 6 or Neigunan), CV8 (Shenque) and ST36 (Zusanli or Stomach 36) are the points. Shenque (CV 8) is centrally located at the midpoint of the umbilicus, with a thin stratum corneum and free of adipose tissue, so application is easy. In addition, the application of pressure to this point with tape is very comfortable as it is an application that the person can do by himself. There are studies showing that tape compression technique used alone on the CV8 point can be used in women's health, digestive and respiratory diseases (Wang and Liu 2013; Xin et al. 2011; Huang and Liu 2013; Wang et al. 2014; Yu et al. 2018; Engin 2021). According to the study published by Wang et al. in 2014, 124 people who experienced nausea and vomiting due to amifostine were randomly divided into two groups. The intervention group consisting of 62 people was asked to stick tapes prepared with ginger on the CV8 points.After the intervention, the incidence of nausea and vomiting in the CV8 group was found to be significantly lower than in the control group (Wang et al. 2014). In a case report published by Engin (2021), in our country, a 5-year-old boy who applied to the pediatric outpatient clinic due to motion sickness was recommended to stick a tape on the P6 and CV8 points. The application was tried on the first trip after the recommendation and it was learned that he did not have any complaints during the 7-hour drive on the road (Engin 2021).

Informing about what to do to reduce or eliminate nausea and vomiting, which is a common problem in early pregnancy, is important in terms of alleviating or eliminating nausea and vomiting and increasing the quality of life of pregnant women. Although there are studies in the literature on general nausea-vomiting and motion sickness in childhood, there is no study examining the effect of band-aid applied to the umbilical area (Shenque-CV8 point) on nausea and vomiting during pregnancy. Therefore, the effect of the Band-Aid applied to the umbilical area (Shenque-CV8 point) on nausea-vomiting during pregnancy is wondered.The aim of this study is to examine the effect of a band-aid applied to the umbilical area on nausea-vomiting during pregnancy. (Shenque-CV8 point)

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* 5-14 weeks pregnant,
* Volunteer to participate in the research
* Having nausea and vomiting during pregnancy,
* Not allergic to any drug or product, literate,
* Can speak and understand Turkish
* Pregnant women who did not receive hyperemesis gravidarum treatment will be included.

Exclusion Criteria:

* pregnant over 14 weeks,
* low risk in pregnancy,
* with chronic disease,
* Having multiple pregnancies.
* In order to ensure the follow-up of the application of the women, the researchers will be in constant communication with the women and will check whether they have applied the Band-Aid.
* Women who do not perform the application although they are in the application group will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Rhodes Nausea and Vomiting Index | time frame : 5 days
  The Rhodes Nausea and Vomiting Index rating system is a five-point Likert type, with the lowest possible score being "8" and the highest score being "40". Those who score 8 or below in the RBMI are evaluated as "No Symptom", those between 9-18 points as "Mild Symptom", those between 19-32 points as "Moderate Symptom" and those between 32-40 points as "Severe/Severe Symptom".
Pregnancy Nausea-Vomiting Severity Evaluation Test (PUQE) | time frame : 5 days
  There are 3 questions in the PUQE test that examine nausea, vomiting and retching, respectively. Although symptoms were initially questioned for the last 12 hours, they were later updated to include the last 24 hours (104). In the study conducted by Sucu et al. on pregnant women in Turkey, they stated that the PUQE test is a suitable tool for evaluating the severity of nausea and vomiting during pregnancy. When evaluating the PUQE test, a total score of 3-6 is indicated as mild, 7-12 as moderate, and 13-15 as severe nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlacı Başkaya, Study Director — Sakarya University
Locations (1):
- Yeni Yalı Aile Sağlığı Merkezi, Köseköy, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laitinen L, Nurmi M, Ellila P, Rautava P, Koivisto M, Polo-Kantola P. Nausea and vomiting of pregnancy: associations with personal history of nausea and affected relatives. Arch Gynecol Obstet. 2020 Oct;302(4):947-955. doi: 10.1007/s00404-020-05683-3. Epub 2020 Jul 11. PMID 32653947
- [Background] Einarson TR, Piwko C, Koren G. Prevalence of nausea and vomiting of pregnancy in the USA: a meta analysis. J Popul Ther Clin Pharmacol. 2013;20(2):e163-70. Epub 2013 Jul 14. PMID 23863545
- [Background] Yu S, Wen Y, Xia W, Yang M, Lv Z, Li X, Li W, Yang S, Hu Y, Liang F, Yang J. Acupoint herbal plaster for patients with primary dysmenorrhea: study protocol for a randomized controlled trial. Trials. 2018 Jul 3;19(1):348. doi: 10.1186/s13063-018-2682-8. PMID 29970155
- [Background] Viljoen E, Visser J, Koen N, Musekiwa A. A systematic review and meta-analysis of the effect and safety of ginger in the treatment of pregnancy-associated nausea and vomiting. Nutr J. 2014 Mar 19;13:20. doi: 10.1186/1475-2891-13-20. PMID 24642205